CLINICAL TRIAL: NCT00587171
Title: A Randomized Trial Comparing Patching With Active Vision Therapy to Patching With Control Vision Therapy as Treatment for Amblyopia in Children 7 to <13 Years Old
Brief Title: Trial Comparing Patching With Active Vision Therapy to Patching With Control Vision Therapy as Treatment for Amblyopia
Acronym: ATS12
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped due to insufficient recruitment.
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-138; 2U10EY011751 (NIH)
Record Dates: First submitted 2007-12-10; First posted 2008-01-07 (Estimated); Results first posted 2011-05-18 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; Vision Therapy; Patching
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): 2 hours of daily patching combined with 1 hour daily of near activities (that includes 30 minutes of at-home active vision therapy) and weekly in-office active vision therapy
  Interventions: Device: Patching; Procedure: Near activities; Procedure: Active vision therapy
- Control (Sham Comparator): 2 hours of daily patching combined with 1 hour of daily near activities (that includes 30 minutes of at-home control vision therapy) and weekly in-office control vision therapy
  Interventions: Device: Patching; Procedure: Near activities; Procedure: Control vision therapy

INTERVENTIONS:
Device: Patching — 2 hours daily patching
  Other Names: Coverlet, 3M Opticlude, Ortopad®
Procedure: Near activities — 30 minutes daily near activities at home
Procedure: Active vision therapy — 30 minutes of daily at-home active vision therapy and a weekly 45 minute in-office active vision therapy session
  Arms: Active
Procedure: Control vision therapy — 30 minutes of daily at-home control vision therapy and a weekly 45 minute in-office control vision therapy session
  Arms: Control

SUMMARY:
This study is comparing the effectiveness of patching combined with active vision therapy plus near activities versus patching combined with control vision therapy plus near activities for moderate amblyopia (20/40-20/100) in 7 to <13 year olds.

The primary outcome measure is the proportion of patients with visual acuity of 20/25 or better in the amblyopic eye at the 17-week masked exam. These patients will be considered treatment responders. The primary analysis will consist of a comparison between the 2 treatment groups of the proportion of treatment responders with adjustment for baseline visual acuity.

Secondary outcomes are stereoacuity at the 17-week masked exam, mean improvement in visual acuity at the 17-week masked exam, and rate of improvement of visual acuity.

DETAILED DESCRIPTION:
Patching and atropine have been traditionally used for the improvement of visual acuity in children with amblyopia. Previous studies have shown that these methods of treatment are effective in young children with functional amblyopia. More recently ATS3, a randomized clinical trial of 507 children ages 7-<18, found that part-time patching combined with atropine and near activities improved visual acuity by two or more lines in 53% of the 7 to 12 year olds compared to 25% for optical correction alone. For the 13 to 17 year olds, part-time patching and near activities improved visual acuity by 2 or more lines in 25%, compared to 23% for optical correction alone. While it appears that patching and/or atropine, combined with near activities, can improve visual acuity in some patients ages 7-<18, most patients in the study were left with residual visual acuity deficits. To further improve visual acuity and binocularity in children with amblyopia some eye care providers augment these traditional therapies with vision therapy. Vision therapy is prescribed initially if there is moderate amblyopia with stereopsis. Vision therapy can be added to the treatment regimen once the patient has reached moderate levels of vision loss with stereopsis and if the patient is still not responding to the current treatment and still has moderate amblyopia. It is thought that the best candidates for this type of therapy are those children with a minimum level of stereopsis (at least 800") and without constant strabismus. Those children with no stereopsis would not be able to perform the activities in the later stages of therapy utilizing binocular vision.

Vision therapy is a sequence of prescribed activities typically performed on a daily basis at home and weekly in-office, and is directed toward an individual patient's deficient skills. Visual skills are practiced under conditions that provide the patient with feedback. The feedback, along with a gradual increase in the demand of the activities as improvement occurs, enables the patient to improve visual functions such as visual acuity, fixation, accommodation, and vergence skills.

There have been case reports and small sample studies that have shown that vision therapy in combination with spectacles and occlusion is effective in improving the visual acuity of patients with amblyopia. Wick et al looked at nineteen patients who were diagnosed with anisometropic amblyopia between the ages of 6 to 49. Seventeen of the patients had moderate amblyopia and two had severe amblyopia, based on the definition of amblyopia used in the Amblyopia Treatment Studies. The patients were treated with a sequence that included spectacle correction, occlusion therapy and both monocular and binocular vision therapy. Thirteen of the seventeen patients with moderate amblyopia had a final visual acuity of 20/25 or better and all of the patients with moderate amblyopia had 20/30 or better final visual acuity.

More recent reports on "perceptual learning," an active form of therapy in which amblyopic subjects practice a position-discrimination task, have shown a mean acuity improvement of approximately 30% (two lines) in amblyopic children and adults who had completed occlusion therapy. These studies provide support for the notion that the practice of particular visual skills under conditions that provide the patient with feedback (e.g., vision therapy) may be beneficial in improving the visual performance of amblyopic eyes.

The second reason to prescribe active therapy is to enhance or facilitate the effects of occlusion by directly treating the aforementioned deficits found to be associated with amblyopia. Most therapy procedures are designed to remediate specific deficiencies in four main areas: fixation, spatial perception, accommodative efficiency, binocular function and oculomotor control.

Lastly, some investigators have suggested that the use of vision therapy may reduce the likelihood of recurrence of the amblyopia. This may be particularly true with anisometropic amblyopia in which vision therapy can be used to improve binocular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 to <13 years
* Amblyopia associated with anisometropia, strabismus (comitant or incomitant), or both at the time of the eligibility examination
* Visual acuity in the amblyopic eye between 49 and 71 letters inclusive (20/40 to 20/100 inclusive) on the eETDRS
* Visual acuity in the sound eye of 79 or more letters on the eETDRS (20/25 or better)
* Inter-eye acuity difference of 15 or more letters (3 or more logMAR lines)
* At least 800 seconds of arc on the Randot Preschool Stereoacuity Test
* Previous or current amblyopia treatment with spectacles or contact lenses, patching or atropine is permitted.
* No myopia more than -6.00 D spherical equivalent in the amblyopic eye
* Single vision spectacles, if needed, worn for at least 16 weeks or until visual acuity documented to be stable
* The child has access to a computer on a daily basis (to use the home vision therapy software)

Exclusion Criteria:

* Previous vision therapy or orthoptics
* Known skin reactions to patch or bandage adhesives
* Prior intraocular or refractive surgery
* Bifocals
* Constant strabismus at near at the eligibility examination
* A family member is (or has been) enrolled in this study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don W. Lyon, O.D., Study Chair — Indiana University; David T. Wheeler, M.D., Study Chair — Casey Eye Institute
Locations (7):
- United States (7):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Bascom Palmer Eye Institute, Miami, Florida
  - Indiana University School of Optometry, Bloomington, Indiana
  - Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Family Eye Group, Lancaster, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee

REFERENCES:
- [Result] Lyon DW, Hopkins K, Chu RH, Tamkins SM, Cotter SA, Melia BM, Holmes JM, Repka MX, Wheeler DT, Sala NA, Dumas J, Silbert DI; Pediatric Eye Disease Investigator Group. Feasibility of a clinical trial of vision therapy for treatment of amblyopia. Optom Vis Sci. 2013 May;90(5):475-81. doi: 10.1097/OPX.0b013e31828def04. PMID 23563444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen subjects were recruited by 7 community based or institutional based sites between April 2008 and March 2009.
Pre-assignment Details: At enrollment, subjects were required to have been treated with at least 16 weeks of single vision spectacles (if needed) or until visual acuity was documented to be stable. The child must have had access to a computer on a daily basis.
Period: Overall Study
Arm/Group | Active | Control
Started | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment in years
  years | 10.1 (2.1) | 10.0 (1.8) | 10.0 (1.9)
Age, Customized [Number; unit: participants] — Age at enrollment in years
  participants
    7 years old | 1 | 2 | 3
    8 years old | 2 | 1 | 3
    9 years old | 2 | 2 | 4
    10 years old | 1 | 0 | 1
    11 years old | 0 | 4 | 4
    12 years old | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 5 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 5 | 8
  Black/African American | 0 | 1 | 1
  Hispanic | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Cause of Amblyopia [Number; unit: participants]
  Anisometropia | 4 | 5 | 9
  Strabismus | 0 | 2 | 2
  Strabismus and anisometropia | 5 | 3 | 8
Distance visual acuity in amblyopic eye [Number; unit: participants] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  participants
    20/100 (48 to 52 letters) (worse) | 2 | 2 | 4
    20/80 (53 to 57 letters) | 0 | 1 | 1
    20/63 (58 to 62 letters) | 1 | 1 | 2
    20/50 (63 to 67 letters) | 4 | 2 | 6
    20/40 (68 to 72 letters) (best) | 2 | 4 | 6
Mean (SD) Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: letters] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  letters | 62.3 (6.8) | 61.9 (7.9) | 62.1 (7.2)
Distance visual acuity in fellow eye [Number; unit: participants] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  participants
    20/40 (68 to 72 letters) (worse) | 0 | 0 | 0
    20/32 (73 to 77 letters) | 0 | 0 | 0
    20/25 (78 to 82 letters) | 2 | 2 | 4
    20/20 (83 to 87 letters) | 4 | 5 | 9
    20/16 (88 to 92 letters) (best) | 3 | 3 | 6
Mean (SD) Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: letters] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  letters | 85.3 (3.6) | 86.2 (4.0) | 85.8 (3.8)
Mean (SD) Intereye Acuity Difference [Mean (Standard Deviation); unit: letters] — The difference between eyes in letters was calculated with positive values indicating sound eye better.
  letters | 23.0 (6.5) | 24.3 (8.8) | 23.7 (7.6)
Randot Preschool stereoacuity [Number; unit: participants] — The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc on patients as young as 2 years of age. This Stereotest is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best) seconds of arc. If two shapes are identified correctly the patient progresses to the next lower stereoacuity level. A failed test occurs when the patient cannot identify any shapes.
  participants
    40 arcsec | 0 | 0 | 0
    60 arcsec | 0 | 0 | 0
    100 arcsec | 2 | 4 | 6
    200 arcsec | 3 | 2 | 5
    400 arcsec | 1 | 2 | 3
    800 arcsec | 3 | 2 | 5
    >800 arcsec | 0 | 0 | 0
    Failed pretest | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Distance Visual Acuity in Amblyopic Eye at 17-week Outcome
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
Time Frame: 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
participants
  20/80 (53 to 57 letters) (worse) | 0 | 1
  20/63 (58 to 62 letters) | 1 | 0
  20/50 (63 to 67 letters) | 0 | 2
  20/40 (68 to 72 letters) | 3 | 1
  20/32 (73 to 77 letters) | 0 | 2
  20/25 (78 to 82 letters) | 2 | 2
  20/20 (83 to 87 letters) (best) | 2 | 1

2. Primary Outcome: Mean (SD): Distance Visual Acuity in Amblyopic Eye at 17-week Outcome
Description: as for outcome 1
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 75.6 (9.7) | 72.0 (9.6)

3. Primary Outcome: Distribution of Change in Amblyopic Eye Visual Acuity From Baseline to 17 Weeks
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. A difference was calculated as the difference in letters between baseline and outcome with positive difference indicating improvement in acuity.
Time Frame: Baseline to 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
participants
  >=1 letter worse | 0 | 0
  0 letters | 0 | 0
  1 to 4 letters better | 0 | 2
  5 to 9 letters better | 4 | 4
  10 to 14 letters better | 1 | 2
  >=15 letters better | 3 | 1

4. Primary Outcome: Mean (SD) of Change in Amblyopic Eye Visual Acuity From Baseline to 17 Weeks
Description: as for outcome 3
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 12.0 (5.3) | 8.8 (5.3)

5. Secondary Outcome: Distribution of Fellow Eye Visual Acuity at 17 Weeks
Description: as for outcome 1
Time Frame: 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
participants
  20/25 (78 to 82 letters) (worse) | 2 | 0
  20/20 (83 to 87 letters) | 1 | 4
  20/16 (88 to 92 letters) | 5 | 2
  20/12 (93 to 97 letters) (best) | 0 | 3

6. Secondary Outcome: Mean (SD) of Fellow Eye Visual Acuity at 17 Weeks
Description: as for outcome 1
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 86.5 (4.1) | 89.8 (3.6)

7. Secondary Outcome: Distribution of Change in Fellow Eye Visual Acuity From Baseline to 17 Weeks
Description: as for outcome 3
Time Frame: Baseline to 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
participants
  Within 4 letters | 7 | 7
  5 to 9 letters better | 1 | 2

8. Secondary Outcome: Mean (SD) of Change in Fellow Eye Visual Acuity From Baseline to 17 Weeks
Description: as for outcome 3
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 0.4 (2.8) | 2.9 (2.7)

9. Secondary Outcome: Mean (SD) of Intereye Visual Acuity at 17 Weeks
Description: as for outcome 1
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 10.9 (9.2) | 17.8 (9.4)

10. Secondary Outcome: Mean (SD) of Change in Intereye Visual Acuity From Baseline to 17 Weeks
Description: as for outcome 3
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
letters | 11.6 (4.2) | 5.9 (5.0)

11. Secondary Outcome: Distribution of Randot Preschool Stereoacuity at 17 Weeks
Description: The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc. This Stereotest is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best) seconds of arc. If two shapes are identified correctly the patient progresses to the next lower stereoacuity level. A failed test occurs when the patient cannot identify any shapes.
Time Frame: 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 9
participants
  40 arcsec (best) | 2 | 1
  60 arcsec | 1 | 0
  100 arcsec | 2 | 1
  200 arcsec | 0 | 4
  400 arcsec | 2 | 0
  800 arcsec | 1 | 1
  >800 arcsec (worse) | 0 | 1
  Failed pretest | 0 | 1

12. Secondary Outcome: Distribution of Change in Randot Preschool Steroacuity From Baseline to 17 Weeks
Description: The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc on patients as young as 2 years of age. This Stereotest is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best) seconds of arc. If two shapes are identified correctly the patient progresses to the next lower stereoacuity level. A failed test occurs when the patient cannot identify any shapes.
Time Frame: Baseline to 17 weeks
Measure: Number; unit: participants
Arm/Group | Active | Control
Number analyzed (Participants) | 8 | 8
participants
  2 or more levels worse | 1 | 2
  Within 1 level | 4 | 4
  2 or more levels better | 3 | 2

ADVERSE EVENTS:
Arm/Group | Active | Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
The study was stopped prior to achieving the goal of 45 subjects enrolled due to slow recruitment, leaving only 19 subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No